CLINICAL TRIAL: NCT05407337
Title: Single Center, Randomized, Comparative, Prospective Interventional Study Evaluating the Impact of Brief Psychotherapy by Narrative Exposure Therapy (NET) on the Reduction of Symptoms of Post Traumatic Stress Disorder in Refugee and Asylum Seeking Women in the Program SINDIANE in Marseille
Brief Title: The Effect of Narrative Exposure Therapy Intervention on Post-traumatic Stress Dissorder and Personal Recovery in Refugees and Asylum Seekers of Sindiane Programme
Acronym: SINDIANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-A01172-39
Record Dates: First submitted 2022-05-23; First posted 2022-06-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Beneficiaries of NET therapy + standard Sindiane program management.
  Interventions: Behavioral: Psychotherapy using Narrative Exposure Therapy (NET)
- Control group (No Intervention): Beneficiaries of the standard care of the Sindiane program.

INTERVENTIONS:
Behavioral: Psychotherapy using Narrative Exposure Therapy (NET) — There are four NET sessions, each lasting thirty minutes and defined in advance on a weekly basis. The first session is the one where the person concerned will establish his/her "Life Line" and start his/her life story with the peer mediator.
  The second and third session will be the one where the person will continue his life story. Each session will begin with the mediator reading the story from the previous session, with the person concerned modifying the story if they wish.
  The fourth session will also start with the reading of the story from the previous session and will finish the story if necessary. It will also be the occasion to give the printed story to the person concerned at the end of the session and have it signed by the mediator and the patient.
  To prevent a possible risk of decompensation of the subject during the session, there will be a psychiatrist on site at the time of the NET to be available if the patient needs it.
  Arms: Experimental group

SUMMARY:
Displaced people, like refugees or asylum seekers, have high rate of potentially traumatic events. PTSD is one of the most common psychiatric trouble in this population. It requires specialized support and psychosocial program. Narrative Exposure Therapy (NET), a german psychotherapy, was developed in the 2000 to specifically treat psycho-trauma in this population. It is brief, effective on complex trauma and can be delivered by trained non-caregivers. All published randomized studies have conclued that NET is effetive, but there are still insifficient numbers to make recomendations. To our knowledge, NET has never been tested in France. In Marseille, SINDIANE is a community support and program for refugees and asylum seekers. Many workshops led by peer workers are offered to increase empowerment of beneficiaries and hel them to recover. The development of a NET workshop would make it possible to combine community support and specific and validated psychotherapy. Through this study, the investigators hypothesize that tratment of PTSD with NET in the community-based SINDIANE program decrease symptoms of PTSD.

DETAILED DESCRIPTION:
Methods and design Forty-six participants with a diagnosis of PTSD disorder within the SINDIANE program will be recruited. A prospective single-blind randomized clinical trial will be conducted comparing two groups, one participant in the classic SINDIANE program and one being treated in addition by NET workshp. The evaluations will be done at the baseline, after the intervention and at three and six months follow-up. IN addition, the qualitative and participatory research method called photovoice will be used to better understand the experiences of participants who recieve NETtroughout their recovery.

The primary objective is the assessment of the symptom intensity score (PCL-5) of posttraumatic stress disorder (PTSD).

Secondary objectives are represented by:

* The assessment of the stability over time of the PTSD symptom intensity score at three months and six months (PCL-5).
* Assessment of the intensity of global psychiatric comorbidities (RHS-15)
* Evaluation of life indicators: ability to act, quality of life (GSE self-efficacy questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18
* Refugee or asylum seeker (habing applied to OFFPRA or with a residence permit)
* Belonging to the SINDIANE community project
* Having been exposed to at least one traumatic event (according to the DSM 5 definition validated by a doctor)
* Having a PCL5 score greater than 23
* Agreeing to participate in the study with an informed consent signed by the subject after explanations given by the investigating psychiatrist
* Patient affiliated to a social security health care
* Patient able to read and write arabic or french

Exclusion Criteria:

* Be under the age of 18
* Be included in another intervention research
* Presence of severe mental retardation or dementia according to DSM5
* Persons benefiting from special protection : under article L3212-1 and L3213-1 of the Public Health Code
* Persons referred to in articles L1121-5 to L1121-8 of the CSP
* Existence of a high suicide risk assessed by the R.U.D.
* Patient subject to a compulsory care measure (Law n°2011-803 of july 5, 2011 relating to the rights and protection of persons subject to psychiatric care and the terms of care)
* Patient refusing to sign the consent or unable to receive the information necessary to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Refugee women aged 18 and over and asylum seekers in the SINDIANE program
Enrollment: 46 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms measure by PCL5 | 1 month post NET therapy
  The PCL-5 is a self reported score. The higher the score, the greater intensity of the symptoms of PTSD. It is validated in english and french with goof psychometric characteristic. The total score of the questionnaire is 80. The scale varies per question from 0 to 4:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely
  If the patient gets a 0, it means that he/she does not have this symptom of post-traumatic stress. On the contrary, the more the score increases and tends towards 4, the more the symptom will be present in the patient.

SECONDARY OUTCOMES:
Evolution of PCL5 score | 3 months and 6 months
  Comparaison of the PCL-5 score after therapy and at 3 and 6 moth. This endpoint is intersted in highlighting a possible improvement in symptoms at a distance from the therapy.
  The total score of the questionnaire is 80. The scale varies per question from 0 to 4:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely
  If the patient gets a 0, it means that he/she does not have this symptom of post-traumatic stress. On the contrary, the more the score increases and tends towards 4, the more the symptom will be present in the patient.
Psychiatric comorbidity intensity score RHS15 | before the intervention, 1 month post therapy, 3 months and 6 months
  Since post traumatic stress disorder is often accompanied by comorbid disorders such as depression or addictive behavior disorder. This evaluation will allow us to assess the possible effectiveness of NET on the associated disorder. This judgment criterion will be assessed using RHS15 wich is a self administrated questionnaire validated in the creening of the main psychiatric disorders.
  The total of the base varies between 0 and 56. By question the scale varies between 0 and 4:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely A score of 0 means that the patient does not have a psychiatric disorder. The higher the score, the more the patient will have more and more mental disorders.
EvExperience indicators intensity score (GSE) | before the intervention, 1 month post therapy, 3 months and 6 months
  This main judgment criterion is concerned with the overall functioning of person concerned. Indeed, it makes it possible to evaluate the satisfaction and the power to act of the person. It is used to have a broader assesment of the expected benefits of PTSD treatment.
  The total score varies between 10 and 40. The more the patient scores, the higher his or her sense of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hôpitaux Marseille; Clotilde IZABELLE, Dr, Principal Investigator — Assistance Publique Hôpitaux Marseille
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, Bouches-du-Rhône, France